CLINICAL TRIAL: NCT05829525
Title: Relationship Between Sleep Quality, Sleep Duration, Heart Rate, and Step Number in Young Adults
Brief Title: Relationship Between Sleep Quality, Sleep Duration, Heart Rate, and Step Number
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 83116987-614
Record Dates: First submitted 2023-03-12; First posted 2023-04-25 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-09

CONDITIONS: Healthy Young Adult
Keywords: Step count; Physical activity; Heart rate; Sleep quality; Sleep duration
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Sleep Duration; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy young adults group (Other): Face-to-face assessment study
  Interventions: Other: Evaluation of sleep quality, sleep duration, heart rate and step count

INTERVENTIONS:
Other: Evaluation of sleep quality, sleep duration, heart rate and step count — Evaluation of sleep quality with the Pittsburgh Sleep Quality Index Evaluation of sleep duration, heart rate, and step count with the Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA) Evaluation of quality of life with the Nottingham Health Profile

SUMMARY:
This study aims to evaluate the relationship among sleep duration, heart rate, number of steps, and sleep quality.

DETAILED DESCRIPTION:
There are studies examining the relationship between sleep quality and physical activity in young adults. In these studies, weakly significant relationships were recorded between sleep quality and physical activity level. However, in these studies, the level of physical activity was evaluated with the International Physical Activity Questionnaire and the questionnaire was filled in within the framework of certain activities. In this study, physical activity will be evaluated with the number of steps taken per day. In addition, there is no study examining the relationship between sleep quality, sleep duration, and heart rate in young adults. With the current study, parameters that will affect physical activity such as sleep duration, heart rate, and the number of steps will be evaluated and their relationship with sleep quality will be determined. Sleep quality will be assessed by the Pittsburgh Sleep Quality Index, sleep duration, heart rate, and step count will be assessed by the Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA), and quality of life will be assessed by the Nottingham Health Profile. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30,
* Without any chronic disease,
* No past or present mental illness,
* Can speak, read, and write Turkish and
* Who volunteered to participate in the study

Exclusion Criteria:

* With any neurological, psychiatric or cognitive impairment,
* Who cannot speak, read or write Turkish

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 1 day
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality. PSQI is a scale that provides information on sleep quality and the type and severity of sleep disturbance in the past week. Turkish validity and reliability were established. In the scale consisting of 24 questions in total, 19 questions are answered by the person, while the other 5 questions are filled by the person's bedmate. 7 sub-dimensions (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are evaluated with 19 questions answered by the individual. Each item in the scale scores between 0 (no distress)-3 (severe distress). The sum of the scores of the seven subdimensions gives the total PSQI score (between 0-21). Those with a total score of 5≥ "good sleep", and those with a score of 5< are considered "poor sleep quality".
Sleep duration | Single assessment for 1 day
  Sleep time will be evaluated with the Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA). Individuals will wear a Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA) on one wrist. During a day, individuals' sleep duration will be recorded. They will be asked to continue with their normal routines, in abnormal cases the measurement will be repeated. Data will be transferred via Bluetooth to smartphones or tablets accessible via the Fitbit App. Individuals' privacy will be protected by downloading the Fitbit app only to the principal investigator's device and creating separate accounts, one for each Fitbit device, without providing personal information.
Nottingham Health Profile | 1 day
  The Nottingham Health Profile (NHP) will be used to assess quality of life. The NHP is a general quality of life questionnaire that measures the perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items. Questions are answered as 'yes' or 'no'. The questionnaire assesses six parameters related to health status. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), emotional reactions (9 items). Each subparameter is scored between 0-100. 0 indicates best health, 100 indicates worst health. The total NHP score is derived from the sum of the subscores.
Heart rate | 1 day
  Heart rate count will be evaluated with the Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA). Individuals will wear a Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA) on one wrist. During a day, individuals' heart rate will be recorded. They will be asked to continue with their normal routines, in abnormal cases the measurement will be repeated. Data will be transferred via Bluetooth to smartphones or tablets accessible via the Fitbit App. Individuals' privacy will be protected by downloading the Fitbit app only to the principal investigator's device and creating separate accounts, one for each Fitbit device, without providing personal information.
Step count | 1 day
  Step count will be evaluated with the Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA). Individuals will wear a Fitbit® Inspire 2 (Fitbit, Inc., San Francisco, California, USA) on one wrist. During a day, individuals' step count will be recorded. They will be asked to continue with their normal routines, in abnormal cases the measurement will be repeated. Data will be transferred via Bluetooth to smartphones or tablets accessible via the Fitbit App. Individuals' privacy will be protected by downloading the Fitbit app only to the principal investigator's device and creating separate accounts, one for each Fitbit device, without providing personal information.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No